CLINICAL TRIAL: NCT02742402
Title: DIAgnostic iMaging or Observation in Early Equivocal appeNDicitis - a Randomized Controlled Trial
Brief Title: DIAgnostic iMaging or Observation in Early Equivocal appeNDicitis
Acronym: DIAMOND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Panu Mentula, M.D., Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUS/95/2016
Record Dates: First submitted 2016-04-07; First posted 2016-04-19 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — X-Rays; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation (Experimental): Clinical follow-up for at least 6-8 hours, after follow-up repeated laboratory tests and repeated clinical examination is done. Adult Appendicitis Score is calculated after observation to determine further actions. Observation is continued in patients with decreasing score. Patients with the same or higher score undergo diagnostic imaging (score 11-15) or laparoscopy (score 16 or higher). Diagnostic imaging is abdominal ultrasound first and if the result is inconclusive or negative for appendicitis abdominal computed tomography is done. Laparoscopic appendectomy is done for those patients with appendicitis in diagnostic imaging.
  Interventions: Other: Observation
- Diagnostic imaging (Active Comparator): Patients undergo abdominal ultrasound and if the result is inconclusive or negative for appendicitis patients will have abdominal computed tomography. Laparoscopic appendectomy is done for patients with appendicitis in diagnostic imaging.
  Interventions: Other: Diagnostic imaging

INTERVENTIONS:
Other: Diagnostic imaging — Abdominal ultrasound, followed by abdominal computed tomography when necessary
  Arms: Diagnostic imaging
Other: Observation — Observation for 6 to 8 hours. After observation period repeated clinical examination and repeated blood test for calculation of Adult Appendicitis Score is done.
  Arms: Observation

SUMMARY:
The aim of the study is to evaluate whether patients with early equivocal appendicitis can be observed instead of immediate diagnostic imaging. Half of the patients are randomly assigned to observation group, while the other half will undergo diagnostic imaging. The hypothesis is that resolving appendicitis is common in these patients. Thus, in observation group there will be fewer patients with appendicitis diagnosis and observation reduces the use of diagnostic imaging and surgery.

DETAILED DESCRIPTION:
For the study equivocal appendicitis is defined as clinical suspicion of appendicitis with Adult Appendicitis Score between 11 and 15. The estimated prevalence of appendicitis in such patients is around 50%.

Diagnostic imaging is done using conditional computed tomography i.e. abdominal ultrasound first and computed tomography only after negative or inconclusive appendicitis after ultrasound.

In observation group repeated clinical examination is done after 6-8 hours interval with repeated blood test for calculation of Adult Appendicitis Score. Patients with decreasing score value continue observation without imaging, whereas patients with the same score value or higher (but below 16) undergo diagnostic imaging as in other group. Laparoscopy is done without imaging in patients with high score (16 or higher). Antibiotics are not allowed, but prophylactic antibiotics during induction of anesthesia are allowed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of acute appendicitis
* Equivocal appendicitis defined by Adult Appendicitis Score: Score ≥11 and ≤15.

Exclusion Criteria:

* C-reactive protein >99 mg/l
* Time from symptom onset over 24 hours
* Pregnancy
* Antibiotics given within last 24 hours
* Suspicion of other disease than appendicitis, that would require immediate interventions such as surgery, diagnostic imaging or gynecologic consultation
* Missing written informed consent
* Patient randomized earlier to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Appendicitis requiring surgery or other intervention | 30 days from randomization

SECONDARY OUTCOMES:
Complicated appendicitis | 30 days from randomization
  Perforated appendicitis or appendiceal abscess
Delayed appendicitis diagnosis | 30 days from randomization
  Diagnosis is delayed if appendicitis is diagnosed later than 24 hours from randomization
Number of diagnostic imaging studies needed | 30 days from randomization and within 1 year after randomization
  Number of abdominal ultrasound and abdominal computed tomography per patient
Appendicitis requiring surgery or other intervention | within 1 year after randomization
Negative appendectomy | 30 days from randomization
  Laparoscopy done for suspected appendicitis, but patient does not have appendicitis
Number of re-admissions to emergency unit | 1 year
  Any reason for re-admission are accounted
Number of other clinically relevant findings | 30 days from randomization
  Findings unrelated to appendicitis
Number of patients requiring of gynecological consultation | 30 days from randomization
  Applicable only in female patients
Time for decision | 30 days from randomization
  The time from randomization to either decision to operate in appendicitis patients or to discharge in non-appendicitis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Panu J Mentula, M.D. Ph.D., Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Meilahti Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sammalkorpi HE, Mentula P, Leppaniemi A. A new adult appendicitis score improves diagnostic accuracy of acute appendicitis--a prospective study. BMC Gastroenterol. 2014 Jun 26;14:114. doi: 10.1186/1471-230X-14-114. PMID 24970111
- [Derived] Lastunen KS, Leppaniemi AK, Mentula PJ. DIAgnostic iMaging or Observation in early equivocal appeNDicitis (DIAMOND): open-label, randomized clinical trial. Br J Surg. 2022 Jun 14;109(7):588-594. doi: 10.1093/bjs/znac120. PMID 35482016
- See also: Original publication of Adult Appendicitis Score — http://bmcgastroenterol.biomedcentral.com/articles/10.1186/1471-230X-14-114
- See also: Online calculator for Adult Appendicitis Score — http://www.appendicitisscore.com/